CLINICAL TRIAL: NCT05285514
Title: Analysis of the Macro-microcirculatory Coupling in the Course of Using the Vasoactive Substances During Anesthesia-resuscitation of Brain-damaged Patients
Brief Title: Macro- and Microcirculation Crosstalk in Brain-damaged Patients Under Anesthesia or in Intensive Care
Acronym: MICRONOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); LMS Polytechnique (Unknown); M3DISIM Inria Université Paris-Saclay (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP211317; 2021-A02375-36 (Other: IDRCB)
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Brain Injury
Keywords: Hemodynamic monitoring; Microcirculation; Macro-microcirculation crosstalk; Vasoactive agents
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brain-damaged patients under anesthesia and requiring the administration of a vasoactive agent: Patients with severe brain injuries over 18 years of age are eligible to participate in this protocol: head trauma, subarachnoid hemorrhage, ischemic or hemorrhagic stroke and requiring the administration of a vasoactive agent as part of routine medical care to restore Cerebral Perfusion pressure (CPP).
  Interventions: Diagnostic Test: Comparison of macro- and microcirculatory parameters

INTERVENTIONS:
Diagnostic Test: Comparison of macro- and microcirculatory parameters — Microcirculation examination using sublingual videomicroscopy, tissue O2 saturation (StO2) by NIRS and transcutaneous CO2 pressure (tcpCO2) monitoring, in conjunction with macrocirculatory parameters measures including cardiac output, arterial pressure and pulsed O2 saturation, in order to establish the relationship between the macrocirculatory changes in blood pressure and cardiac output and the microcirculatory flow and capillary density during vasoactive agent use." . Participants receive interventions as part of routine medical care to restore Cerebral Perfusion pressure (CPP) to appropriate levels (60-70 mmHg)

SUMMARY:
In patients with severe brain injury, maintenance and control of blood pressure is at the very first point in the management strategy, whether in anesthesia or in intensive care. In order to restore cerebral perfusion pressure (CPP) to appropriate levels (60-70 mmHg) while ensuring optimal perfusion of other vital organs, intravenous administration of vasodilator, inodilator or vasoconstrictor vasoactive agents is commonly used.

These vasoactive agents, widely used to correct hypotension or hypertension, have their own effects on the load conditions of the left ventricle and the tone of the arterial tree, but also have effects on the microcirculation.

The microcirculatory status of a tissue cannot be reliably predicted by considering only the macrocirculatory parameters usually measured.

Therefore, in situations where organ perfusion is inadequate or compromised, patient management that includes the integration of the impact of vasoactive agents on the microcirculation seems essential for comprehensive hemodynamic treatment.

The non-invasive study of microcirculatory perfusion and its interactions with the macrocirculatory network, using a minimally invasive method such as videomicroscopy, should allow a better use of the treatments used.

For cerebral patients, routine management already includes very complete monitoring of all cardiopulmonary and cerebral systemic parameters.

It is therefore imperative to study and propose new minimally invasive modalities for monitoring the microcirculation in order to define new therapeutic targets that take into account the microcirculatory compartment.

DETAILED DESCRIPTION:
In patients with severe brain injury, maintenance and control of blood pressure is at the primary focus of the management strategy in both anesthesia and intensive care. In order to restore cerebral perfusion pressure (CPP) to appropriate levels (60-70 mmHg) while ensuring optimal perfusion of other vital organs, intravenous administration of vasodilator, ino-dilator or vasoconstrictor agents is widely used.

These vasoactive agents widely used to correct hypotension or hypertension have their own effects on left ventricular loading conditions, arterial tree tone, but also effects on microcirculation.

Currently, the vast majority of anaesthesias and organ resuscitations are carried out from a macrocirculatory view of the system. Hemodynamic optimization is then based on the monitoring of macrocirculatory parameters such as arterial pressure, and sometimes cardiac output coupled with parameters of adequacy of tissue oxygenation (arterial and venous O2 saturation).

The microcirculatory status of a tissue cannot be reliably predicted by considering only the usually measured macrocirculatory parameters. Peripheral capillary perfusion pressure is the result of the coupling between peripheral microcirculatory tone and resistance and macrocirculatory impedance.

The response of microvessels to the various vasoactive agents widely used in the clinic has been little studied.

However, it should be noted that excessive use of vasoconstrictor amines, particularly in the presence of hypovolemia, may, paradoxically to the macrocirculatory impression, induce closure of the capillary network and aggravate tissue ischemia. This capillary de-recruitment is due in particular to the dissipation of pressure in the systemic arterial system, due to the excessively high peripheral resistances and fatally leads to a rarefaction of the open capillaries.

In addition, the increased macrocirculatory impedance imposes a myocardial workload that may cause a decrease in cardiac output, amplifying the tissue damage. This leads to a new situation of uncoupling, characterized by decreased macrocirculatory flow and elevated microcirculatory resistance.

This is why, in situations where organ perfusion is inadequate or weakened, patient management that includes the integration of the impact of vasoactive agents on the microcirculation seems essential for global hemodynamic treatment.

Impaired microcirculation is a key pathophysiological factor in organ failure and death in patients. The impact of organ failure (renal, respiratory, cardiac, etc.) on the quality of cerebral oxygenation is major and conditions the brain's recovery potential. Organ failure by its repercussions on the conditions of brain recovery severely worsens the prognosis of brain damaged patients (secondary brain insults of systemic origin (SBISOs)

In order to recognize and avoid the pitfalls associated with these aortocapillary uncoupling mechanisms, specific monitoring of microcirculatory flow and tissue perfusion during the administration of vasoactive agents is largely relevant. The major obstacle is the difficulty of studying microcirculatory behavior at the bedside in a non or minimally invasive manner.

Direct visualization of the capillary circulation in vivo is now possible using a minimally invasive technique of orthogonal spectral polarization (OSP) videomicroscopy and, more recently, Sidestream Dark Field imaging (SDF).

This last technique, validated in humans mainly in septic shock situations, uses a polarized light source whose absorbance by hemoglobin and reflection by other tissues allows the construction of a contrasted image. This technique allows the visualization of capillary networks on the surface of solid organs covered with a thin epithelial layer to a depth of about 300 µm. An analysis of the recorded image assisted by calculation software allows the semi-quantitative calculation of capillary density (proportion of perfused vessels; PPVSL), capillary flow (Microcirculatory Flow Index; MFISL) and heterogeneity (heterogeneity index; HETSL) of these.

To date, several non-invasive techniques are available, each measuring different parameters specific to this microcirculation:

Capillary density, capillary or tissue flow estimation, hemoglobin saturation, oxygenation and tissue CO2 pressure measurements.

The non-invasive study of microcirculatory perfusion and its interactions with the macrocirculatory network, thanks to a minimally invasive method such as videomicroscopy, should allow a better use of the treatments used.

Overall, the trend in anaesthesia and intensive care is increasingly towards individualized management, and the use of monitoring (macro- and microcirculatory) associated with a thorough knowledge of the treatments used (vasoconstrictors, vasodilators and vascular filling in particular) seems to be an essential basis for these considerations.

The empirical use of vasoactive agents, without specific monitoring of these effects, and the unpredictable impact of changes in one of the two compartments on the final state of the system during adequate macrocirculatory resuscitation could even be deleterious at the microcirculatory level.

These pathophysiological concepts specific to macro/microcirculation cross-talk demonstrate the imperative of developing monitoring specific to the microvascular network in critical patients.

The techniques have evolved and the tools are now available and can be used safely in patients.

For brain-damaged patients, routine management already includes a very complete monitoring including all systemic cardio-pulmonary and cerebral parameters. Participants receive interventions as part of routine medical care to restore Cerebral Perfusion pressure (CPP) to appropriate levels (60-70 mmHg)

The availability of minimally invasive monitoring tools of the microcirculation such as videomicroscopy allows the study of the functional capillary situation according to the vasoactive agent used.

The study of microcirculatory perfusion and its interactions with the macrocirculatory network, using a minimally invasive method such as videomicroscopy, should allow a better use of the treatments used.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* With brain damage
* Benefiting from general anesthesia or resuscitation justifying the placement of an arterial catheter and monitoring of cardiac output
* With hypotension or arterial hypertension requiring intravenous administration of a vasoactive agent to meet the target cerebral perfusion pressure (CPP) of 60-70 mmHg
* Not subject to a measure of legal protection (tutorship/curatorship)
* Patients informed and having expressed their non-objection to participation in this research, or, where applicable, a person of trust / family member / relative of the patient who is unable to express her or his agreement

Exclusion Criteria:

* Patients under the age of 18
* Pregnant woman
* Patient without affiliation to a social security scheme
* Patient, or, where applicable, person of trust / family member / relative of the patient unable to express her or his agreement, opposed to participation in the study
* Patient subject to a legal protection measure
* Patient benefiting from the State medical assistance (AME) program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years old) with brain damage, undergoing general anesthesia or intensive care justifying, due to their severity, monitoring of blood pressure and cardiac output.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Capillary density | Duration of the surgical intervention (1 day)
  For all patients, Capillary density by sublingual video microscopy (proportion of perfused vessels; PPVSL / percentage and the heterogeneity index; HETSL / H-unit) will be collected in separate time periods:
  1. Baseline before administration of the vasoactive agent
  2. After 5 minutes
  3. After stabilization 15 minutes
Microcirculatory flow | Duration of the surgical intervention (1 day)
  For all patients, Capillary flow estimation using sublingual videomicroscopy (Microcirculatory Flow Index MFISL/ unit FI) will be collected in separate time periods:
  1. Baseline before administration of the vasoactive agent
  2. After 5 minutes
  3. After stabilization 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Study Director — AP-HP, Lariboisière Hospital, Department of Anesthesiology and Intensive Care; Fabrice VALLEE, MD, PhD, Principal Investigator — AP-HP, Lariboisière Hospital, Department of Anesthesiology and Intensive Care
Locations (1):
- AP-HP, Lariboisière Hospital, Department of Anesthesiology and Intensive Care, Paris, France